CLINICAL TRIAL: NCT07080593
Title: Testing of an Innovative Patient-Centered Physical Activity Program for Hemodialysis Patients
Brief Title: Patient-Centered Physical Activity Program for Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Principal Investigator, Kenneth Wilund, Director of the School of Nutritional Science and Wellness, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21005
Record Dates: First submitted 2021-04-21; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; Physical Activity; Fatigue; Patient Reported Outcomes; Wellness
MeSH Terms: conditions — Motor Activity; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Novel Physical Activity Group (Experimental): The novel PA program included 2 phases, a structured phase and a self-directed phase. During the structured phase, the primary goal was to increase PA levels. Participants had autonomy in selecting their preferred activities, including supervised intradialytic exercises (e.g., cycling or resistance training); at-home exercise (e.g., aerobic, resistance, balance, and flexibility exercises), and lifestyle activities (e.g., gardening, household chores, walking, etc.). Participants were encouraged to progress their PA over time by gradually increasing exercise duration or intensity. During this phase, participants were met with during each dialysis session as scheduling allowed.
  During the self-directed phase. the primary goal was to encourage continued PA by promoting greater participant autonomy. Participants determined the frequency of their visits and goal-setting meetings with the research staff, but were met with at least once per week.
  Interventions: Behavioral: Novel Physical Activity Program
- Standard of care physical activity group (Active Comparator): The standard of care PA program aimed to promote engagement in PA during dialysis treatments, similar to the structure of previous studies14,17,19,20,23. Participants in the comparator group were offered a host of supervised intradialytic exercises, including cycling (Monark information), and 4 resistance exercises: knee flexion, knee extension, calf raises, and seated marching. Participants were met with during each dialysis treatment (approximately 3 times per week, as scheduling allowed) throughout the entire study period to ensure exercises were performed correctly and support progression as appropriate. Participants were encouraged to progress as tolerated. Progression strategies included increasing resistance or exercise duration.
  Interventions: Behavioral: Standard of Care Physical Activity Program

INTERVENTIONS:
Behavioral: Novel Physical Activity Program — A structured phase and a self-directed phase, involving both in center and out-of-center exercise. Our novel intervention provides patient's the autonomy to choose the types of physical activity and exercise that they are willing and able to participate in. In brief, it involves working one-on-one with patients to develop an activity prescription that aligns with the participants' goals and motivations to increase physical activity levels.
  Arms: Novel Physical Activity Group
Behavioral: Standard of Care Physical Activity Program — Those in the control group will undergo a variety of exercises including intradialytic cycling and resistance ("strength training")
  Arms: Standard of care physical activity group

SUMMARY:
Individuals undergoing HD generally have very low physical activity levels, which consequently contributes to elevated levels of perceptions of fatigue, poor physical function, and a decline in overall quality of life, all of which are linked to progressively greater risk for comorbidities and mortality. The various benefits of physical activity for the general population are well understood, showing a dose-response relationship between physical activity and health. While CKD is not reversible, exercise is often encouraged for its potential to slow disease progression, reduce symptom burden, and improve transplant readiness for HD patients. Over the last two decades, efforts have been made to increase physical activity levels in HD patients, yet the benefits are inconsistent and limited. Many interventions have implemented physical activity programs that include simplistic exercise prescriptions, including intradialytic cycling and/or light resistance exercises. These general, non-personalized exercise programs are associated with poor adherence, high dropout rates, and conflicting effects on physical function or other outcomes related to quality of life. As such, many have discussed the need for individualized exercise prescriptions to overcome the barriers that prevent HD patients from meeting national guidelines for exercise.

In this context, the purpose of this study is to compare the efficacy of a personalized, novel intervention (intervention) compared to a standard of care intervention (comparator), and its effect on perceptions of fatigue, self-reported depression, and physical function. Our primary hypothesis is that the intervention group will elicit greater improvement in physical activity levels than the comparator group. Our secondary hypothesis is that the intervention group will elicit greater improvements in perceptions of fatigue, self-reported depression, and physical function than the comparator group.

DETAILED DESCRIPTION:
We have designed a novel physical activity intervention that is designed to overcome many of the barriers to increasing physical activity in this population. The novel physical activity program (intervention group) included 2 phases, a structured phase and a self-directed phase. During the structured phase (weeks 0 through 11), the primary goal was to increase physical activity levels. During the self-directed phase (weeks 13 through 24), the primary goal was to encourage continued physical activity by promoting greater participant autonomy.

The rationale for this approach is that participants are able to choose activities that are important to them, as opposed to prescribed mandated exercises they may not value or benefit from. In brief, it involves working one-on-one with patients to develop an activity prescription that aims to increase the participants' physical activity levels in a sustainable way. Participants had autonomy in selecting their preferred activities, including supervised intradialytic exercises (e.g., cycling or resistance training); at-home exercise (e.g., aerobic, resistance, balance, and flexibility exercises), and lifestyle activities (e.g., gardening, household chores, walking, etc.). This contrasts with what is normally done, which is to assign specific types of exercise that they may not be motivated or willing to do.

If randomized into the control group, this standard of care group aimed to promote engagement in PA during dialysis treatments, similar to the structure of previous studies. Participants in the comparator group were offered a host of supervised intradialytic exercises, including cycling, and 4 resistance exercises: knee flexion, knee extension, calf raises, and seated marching. Participants were met with during each dialysis treatment (approximately 3 times per week, as scheduling allowed) throughout the entire study period t and support progression were encouraged to progress as tolerated.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old (no upper age limit);
* Chronic hemodialysis for ≥ 3 months;
* No planned or expected change in dialysis modality, elective surgery, or relocation during the study period (24 weeks);
* Able to communicate in English or Spanish and provide written informed consent;
* Assessed to be safe and able to exercise by the Hemodialysis unit nephrologist

Exclusion Criteria:

* Physical Activity: patients currently participating in prescribed exercise.
* Physician Clearance: Patients who do not receive physician clearance to participate in the study will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity Levels | Week 0, week 11, week 23
  MET minutes (physical activity time and intensity) based on the 2011 Compendium of Physical Activities.

SECONDARY OUTCOMES:
Change in Fatigue | Week 0, week 11, week 23
  SONG-HD Fatigue measure. Scores range from 0 to 9 with higher scores reflecting greater fatigue.
Change in Depressive symptoms | Week 0, week 11, week 23
  Patient Reported Outcomes Measurement Information System- Depression Short Form 8a
Change in Physical function | Week 0, week 11, week 23
  Short Physical Performance Battery

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wilund, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (3):
- United States (3):
  - US Renal Care, Bolingbrook, Illinois
  - US Renal Care, Oak Brook, Illinois
  - Champaign-Urbana Dialysis Center, Urbana, Illinois

IPD SHARING:
Plan to Share IPD: No